CLINICAL TRIAL: NCT07347353
Title: Molecular HistoMx Assessment for Kidney Transplant Rejection and Management
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: Molecular_kidney rejection
Record Dates: First submitted 2025-12-16; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Graft Rejection
Keywords: molecular diagnosis; kidney transplantation; graft rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — kidney graft biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant recipients from two referral academic center were enrolled in the study
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Transcriptomic analysis of kidney biopsies has demonstrated the potential to improve diagnosis of graft rejection. Molecular assessment of kidney graft rejection based on the Banff Human Organ Transplant consensus gene panel is an available and validated tool (HistoMx). However the applicability of molecular assessment of graft biopsy in real life setting is unclear. The main objective is to assess the clinical need of molecular assessment of kidney graft biopsy for diagnosis in real world clinical practice. The secondary objectives are to measure : clinical outcomes at 12-months follow up including patient survival, graft function and graft survival, diagnosis of graft rejection after integrating molecular assessment to standard histology, biology and immunology, and to evaluate therapeutic changes and impact on clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Kidney recipients older than 18 years of age
* Patients receiving a kidney transplant from a living or brain-dead donor

Exclusion Criteria:

* Patients who have received a previous transplant with an organ other than the kidney
* Patients without available graft biopsy material for molecular HistoMx testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients from two French referral centers
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with molecular assessment of kidney graft biopsy for diagnosis in real world clinical practice | 12 months
  The main objective is to assess the clinical indication and rate of participants with molecular assessment of kidney graft biopsy for diagnosis in real world clinical practice

SECONDARY OUTCOMES:
Graft function at 12 months after graft biopsy | 12 months
  The secondary objectives are to graft function at 12 months after graft biopsy using estimated Glomerular Filtration Rate (eGFR)

OTHER OUTCOMES:
Probability of graft survival after graft biopsy | 12 months
  The objective is to measure probability of graft survival post graft biopsy using the iBox predictive system
Rate of participants with graft rejection diagnosis based on molecular assessment of graft biopsy | 12 months
  The objective is to measure the rate of participants with diagnosis of graft rejection based on molecular assessment
Rate of participants with therapeutic changes based on graft rejection diagnosis | 12 months
  The objective is to measure rate of participants with therapeutic changes based on graft rejection diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Lefaucheur, Principal Investigator — Paris Translational Research Center for Organ Transplantation; Alexandre Loupy, Principal Investigator — Paris Translational Research Center for Organ Transplantation
Locations (2):
- France (2):
  - Paris Bichat university hospital, Paris
  - Paris Saint Louis University hospital, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giarraputo A, Goutaudier V, Robin B, Angelini A, Sablik M, Aubert O, Rosales IA, Smith RN, Roufosse C, Adam B, Haas M, Colvin RB, Lefaucheur C, Mengel M, Zielinski D, Loupy A. Relevance of the Banff Human Organ Transplant Consensus Gene Panel for Detecting Antibody and T-Cell-Mediated Rejection of Kidney Allografts. Kidney Int Rep. 2024 May 4;9(7):2290-2294. doi: 10.1016/j.ekir.2024.04.054. eCollection 2024 Jul. No abstract available. PMID 39081730
- [Background] Zielinski D, Goutaudier V, Sablik M, Divard G, Aubert O, Piedrafita A, Mezine F, Dagobert J, Certain A, Robin B, Gueguen J, Rabant M, Duong van Huyen JP, Sannier A, Randoux-Lebrun C, Maanaoui M, Lionet A, Gibier JB, Gnemmi V, Le Quintrec M, Chauveau B, Vermorel A, Couzi L, Bestard O, Elias M, Louis K, Rosales IA, Smith RN, Kung VL, Anglicheau D, Legendre C, Del Bello A, Huang E, Adam B, Kamar N, Colvin RB, Mengel M, Lefaucheur C, Loupy A. Molecular diagnosis of kidney allograft rejection based on the Banff Human Organ Transplant gene panel: A multicenter international study. Am J Transplant. 2025 Aug;25(8):1631-1642. doi: 10.1016/j.ajt.2025.04.025. Epub 2025 May 8. PMID 40345499